CLINICAL TRIAL: NCT01194063
Title: Use of Omegaven for Parenteral Nutrition Associated Liver Disease
Brief Title: Use of Omegaven Fish Oil Emulsion for Parenteral Nutrition Associated Liver Disease in Infants and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kapiolani Medical Center For Women & Children (Other)
Responsible Party: Principal Investigator, Lynn M. Iwamoto, MD, Associate Professor of Pediatrics, Kapiolani Medical Center For Women & Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107954
Record Dates: First submitted 2010-06-17; First posted 2010-09-02 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cholestasis
Keywords: short bowel syndrome; parenteral nutrition associated liver disease; pediatric
MeSH Terms: conditions — Cholestasis; Short Bowel Syndrome | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omegaven (Experimental): Administration of intravenous Omega-3 fish oil lipid emulsion 1 g/kg continuous infusion over 12-24 hrs
  Interventions: Drug: Omega-3 fish oil lipid emulsion

INTERVENTIONS:
Drug: Omega-3 fish oil lipid emulsion — daily intravenous administration of Omegaven fish oil emulsion
  Other Names: Omegaven

SUMMARY:
Use of a fish oil emulsion to decrease liver disease due to long term intravenous nutrition.

DETAILED DESCRIPTION:
Unlike conventional intravenous fat emulsions, Omegaven™ is comprised solely of fish oils containing primarily omega-3 fatty acids. Animal studies have shown that IV fat emulsions such as fish oil that are high in eicosapentaenic and docosahexaenoic acids reduce impairment of bile flow as seen in cholestasis caused by conventional fat emulsions. It is thought that by administering Omegaven™ in place of conventional phytosterol/soybean fat emulsions, cholestasis may be prevented or reversed, and patients will be able to be maintained on adequate PN for growth until they are able to ingest adequate nutrition enterally. Ongoing studies are addressing safety and efficacy of Omegaven™ in the pediatric population. In this trial, infants and children with parenteral nutrition associated liver disease will receive Omegaven™ as compassionate use to potentially prevent progression of disease. Safety and efficacy are monitored.

ELIGIBILITY:
Inclusion Criteria:

* direct bilirubin > 2 mg/dl x2 consecutive
* parenteral nutrition dependent, expected to continue for at least another 30 days from the first day
* patient must have utilized standard therapies to prevent the progression of liver disease

Exclusion Criteria:

* other primary cause of liver disease not parenteral nutrition-associated
* weight <3 kg
* infant or child enrolled in other clinical trial involving an investigational agent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10-20 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
improving cholestasis | One month, 2 months, 3 months after starting omegaven and 1 month after completing treatment
  decline in serum direct bilirubin levels below 2 cm on 2 serial measures

SECONDARY OUTCOMES:
improving liver function tests | 1 year
  includes ALT, AST, GGT, and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Iwamoto, MD, Principal Investigator — Kapiolani Medical Center For Women & Children
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee SI, Valim C, Johnston P, Le HD, Meisel J, Arsenault DA, Gura KM, Puder M. Impact of fish oil-based lipid emulsion on serum triglyceride, bilirubin, and albumin levels in children with parenteral nutrition-associated liver disease. Pediatr Res. 2009 Dec;66(6):698-703. doi: 10.1203/PDR.0b013e3181bbdf2b. PMID 19687773
- [Background] de Meijer VE, Le HD, Meisel JA, Gura KM, Puder M. Parenteral fish oil as monotherapy prevents essential fatty acid deficiency in parenteral nutrition-dependent patients. J Pediatr Gastroenterol Nutr. 2010 Feb;50(2):212-8. doi: 10.1097/MPG.0b013e3181bbf51e. PMID 20038849